CLINICAL TRIAL: NCT06669936
Title: Efficacy Fo Oral Capsule FMT Combined with Bezlotoxumab Following Initial Failure of FMT Alone
Brief Title: Rescue FMT with Bezlotoxumab for Recurrent C. Difficile Infection
Acronym: ZINFMT
Status: Completed | Type: Observational
Sponsor: Alexander Khoruts (Other)
Responsible Party: Sponsor-Investigator, Alexander Khoruts, PI, University of Minnesota
Organization: University of Minnesota (Other)
Other Study IDs: FMTZinplava001
Record Dates: First submitted 2024-07-22; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-07

CONDITIONS: Recurrent C. Difficile Infection
MeSH Terms: interventions — Fecal Microbiota Transplantation; bezlotoxumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Zinplava/FMT: Patients with recurrent C. difficile infections, who failed FMT. This cohort includes patients treated with a combination of bezlotoxumab (Zinplava) and 2nd FMT.
  Interventions: Drug: Fecal microbiota transplantation ± bezlotoxumab

INTERVENTIONS:
Drug: Fecal microbiota transplantation ± bezlotoxumab — Co-administration of bezlotoxumab and FMT in patients with recurrent C. difficile infections who failed FMT alone.
  Other Names: FMT; Zinplava

SUMMARY:
The goal is to evaluate the benefit of adding bezlotoxumab to repeat fecal microbiota transplantation (FMT) in patients with recurrent Clostridioides difficile infections after failure of FMT alone.

DETAILED DESCRIPTION:
Initial failure of FMT in breaking the cycle of recurrent C. difficile infections is associated with a greater risk of subsequent failure. Previous analysis showed that FMT failure is associated with delayed repair of fecal microbiota at one week after administration. The hypothesis underlying this trial is that increased symptom-free interval by administration of bezlotoxumab can improve the outcomes of a second FMT.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Diagnosis of recurrent C. difficile infection based on symptoms and laboratory confirmation.
3. Failure of standard antibiotic therapies prior to the initial FMT

Exclusion Criteria:

1. Pregnancy.
2. Class III or above heart failure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of recurrent C. difficile infection who suffered a relapse without a new antibiotic provocation within 90 days of FMT.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Clinical failure | 90 days
  Recurrence of C. difficile infection as documented by worsened diarrhea symptoms and laboratory evidence for C. difficile infection in stool.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
All relevant data are going to be published.